CLINICAL TRIAL: NCT02671643
Title: To Determine the Measurement Properties of the ACT in an African American Adolescent Population With Persistent Asthma Followed at a Subspecialty Clinic
Brief Title: To Determine the Measurement Properties of the ACT in an African American Adolescent Population With Persistent Asthma
Acronym: ACT AA
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Academy of Allergy, Asthma, and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1532
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: To determine the measurement properties of the asthma control test (ACT) in a prospective clinical study in an African American adolescent population.

DETAILED DESCRIPTION:
African Americans have a higher rate of asthma (11.2%) compared to whites (7.7%), according to the Centers for Disease Control and Prevention, and this asthma is disproportionally not well-controlled. African Americans have higher mortality from and healthcare utilization for their asthma. Their asthma severity is more likely to be underestimated by their "main asthma provider". African-American adolescents are at particularly high risk of asthma-related morbidity and mortality.

Because asthma control is now the focus of asthma care, assessment of control is the critical step in appropriate management. The two domains of asthma control, impairment and risk, evaluate the role asthma plays in a patient's quality of life and functional capacity on an ongoing basis and the risk their asthma presents for future adverse events. Although NAEPP guidelines contain a rubric for asthma control based on these domains, thus representing the "gold standard" for asthma care, their utilization may be time-consuming and cumbersome to implement in primary care offices, and primary care providers may be unfamiliar with their use. Minorities see subspecialists less often than Caucasians (28.3% vs 41%, p=0.001), and this difference could not be explained by age, gender, health insurance, education, employment, patient preference, or frequency of respiratory symptoms. For primary care practices following these patients, it remains imperative that the tools being used to gauge asthma control be evaluated and validated in this at-risk population.

At this time, there are approximately 17 questionnaires available for use in the assessment of asthma control, although most are not well validated. Of these, the most widely validated and most commonly used instrument is the Asthma Control Test (ACT). The ACT is a self-administered questionnaire intended to assess the impairment domain over the past four weeks and is completed by patients starting at age 12. The ACT has five questions with an overall best score of 25. For primarily adult Caucasian populations, the ACT has been found to be a valid, reliable, and responsive instrument of asthma control, and cut-offs for controlled and not well-controlled asthma (< 19) as well as minimal clinically important (MIC) differences (3 points) have been identified. However, measurement properties of the ACT are lacking in the African American adolescent asthma population. The landmark validation study for the ACT by Schatz et al was comprised of a large sample size of over 300 patients that showed that a cut-off score of 19 as distinguishing well-controlled versus not well-controlled asthmatics. However, the mean age was 35 for that study population, and concerns have been raised as to whether this cut-off is appropriate for adolescents in general. Moreover, concerns have been raised as to the application of these cut-offs for different ethnic populations. Recent studies examining the ACT in pediatric adolescent populations have found higher optimal cut points to distinguish control classifications; these groups included both European cohorts as well as children of Mexican descent in Southern California. The ACT has not been validated in a more ethnically diverse population such as in African American adolescents.

The measurement properties of validity, reliability, and responsiveness are critical to the usefulness of any questionnaire in both clinical and research settings. To date, we have been unable to identify a study that evaluated the measurement properties of the ACT in this at-risk minority population.

Lung function measures are included in the rubric of assessing asthma control by the NAEPP. Per these recommendations, spirometry should be available to physicians caring for asthma patients and used with initiation of treatment, change in asthma control, and every one to two years. While subspecialists often have access to spirometry, office-based spirometry is time-consuming, requires technical ability and staff training, equipment maintenance and calibration, and is not always available or feasible for use in primary care physician offices. Because spirometry may be of limited accessibility to primary care providers, questionnaires are quickly taking a leading role in asthma management. However, African Americans perceive asthma symptoms differently than Caucasians. They report less nighttime awakening and dyspnea, two symptoms that account for 20% of the ACT score, and children are less accurate describing their perceived asthma control. This type of under-reporting reflects a false level of asthma control when queried by the ACT and leads to inappropriate medical management when spirometry is not utilized.

Additionally, health literacy is often underestimated. In a review by Diette of approximately 500 mostly African American patients who were asked to read asthma information, only 27% were able to read at a high school level, the level at which most health information and instructions are written. Patients with limited health literacy and chronic illness know less about how to manage their disease and have a higher likelihood of poorly controlled disease and health status compared to their counterparts with higher health literacy. Due to this, the IOM identifies health literacy as being fundamental to quality care and also considers it a priority in health-care quality and disease prevention. Because currently used questionnaires are often provided to patients at the time of intake at a clinic visit for self-administration, a high level of health literacy in this minority adolescent population is a dangerous assumption that must be considered when addressing the utilization of tools in the assessment of asthma control by primary care providers and subspecialists alike.

As exploratory endpoints, we will obtain fractional exhaled nitric oxide (FeNO) measurements shortly after spirometry is performed. Elevated FeNO indicates eosinophilic airway inflammation and assists in assigning the correct asthma phenotype, which can have implications for asthma management. We will also obtain nasal epithelial lining fluid (ELF) for collection of nasal cytokines and chemokines. This information is useful for expanding our current understanding of the inflammatory mediators involved in asthma-associated airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as African-American
* Ages 12-18 years
* Live within convenient driving distance of the NC Children's Specialty Clinic in Raleigh, NC.
* Physician-diagnosis of persistent asthma
* Current treatment with appropriate therapy for persistent asthma symptoms as per the NHLBI guidelines including: Daily controller medication use for asthma requiring at least low-dose inhaled corticosteroids (ICS). Asthma may range from mild persistent through severe persistent asthma, to include subjects that may require daily or every other day oral corticosteroids for control of asthma symptoms

Exclusion Criteria:

* Children younger than age 12 and older than 18
* Children unable to perform spirometry
* Medical history or underlying health problems that may preclude participation in the protocol per the study physician (including but not limited to cystic fibrosis, chronic bronchitis, recurrent pneumonia, immunodeficiency, hematologic disorders)
* Subjects and families unwilling to travel to the clinic for the required 2 visits
* Other uncontrolled health problems
* Non-English speaking subjects

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 80 African-American adolescents ages 12-18 with a physician diagnosis of persistent asthma. These adolescents are followed at the UNC Asthma Clinic seen by either pediatric pulmonologists or allergists.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04-13 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Cohen's kappa | Baseline Visit
  To determine the agreement of the ACT score at the standard cutpoint of >19 with physician assessment of control using Cohen's kappa.

SECONDARY OUTCOMES:
Sensitivity of ACT Questionnaire | Six Weeks (Follow Up Visit)
  A receiver-operating curve will be used to determine the best ACT cutpoint for assessment of control in this population. A logistic regression model will be used with 'control by physician' as the dependent variable and 'ACT score' as the independent variable. The model will include adjustment for repeated measures (baseline and 6 week visit).

OTHER OUTCOMES:
Specificity of ACT Questionnaire | Six Weeks (Follow Up Visit)
  A receiver-operating curve will be used to determine the best ACT cutpoint for assessment of control in this population. A logistic regression model will be used with 'control by physician' as the dependent variable and 'ACT score' as the independent variable. The model will include adjustment for repeated measures (baseline and 6 week visit).
Cohen's kappa | Six Weeks (Follow Up Visit)
  To determine the agreement of the ACT score at the standard cutpoint of >19 with physician assessment of control using Cohen's kappa.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina
  - NC Children's Specialty Clinic, 4414 Lake Boone Trail, Suite 505, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monzon ME, Manzanares D, Schmid N, Casalino-Matsuda SM, Forteza RM. Hyaluronidase expression and activity is regulated by pro-inflammatory cytokines in human airway epithelial cells. Am J Respir Cell Mol Biol. 2008 Sep;39(3):289-95. doi: 10.1165/rcmb.2007-0361OC. Epub 2008 Apr 3. PMID 18390475
- [Background] Krishnan JA, Diette GB, Skinner EA, Clark BD, Steinwachs D, Wu AW. Race and sex differences in consistency of care with national asthma guidelines in managed care organizations. Arch Intern Med. 2001 Jul 9;161(13):1660-8. doi: 10.1001/archinte.161.13.1660. PMID 11434799
- [Background] Zoratti EM, Havstad S, Rodriguez J, Robens-Paradise Y, Lafata JE, McCarthy B. Health service use by African Americans and Caucasians with asthma in a managed care setting. Am J Respir Crit Care Med. 1998 Aug;158(2):371-7. doi: 10.1164/ajrccm.158.2.9608039. PMID 9700109
- [Background] Cloutier MM, Schatz M, Castro M, Clark N, Kelly HW, Mangione-Smith R, Sheller J, Sorkness C, Stoloff S, Gergen P. Asthma outcomes: composite scores of asthma control. J Allergy Clin Immunol. 2012 Mar;129(3 Suppl):S24-33. doi: 10.1016/j.jaci.2011.12.980. PMID 22386507
- [Background] Juniper EF, Gruffydd-Jones K, Ward S, Svensson K. Asthma Control Questionnaire in children: validation, measurement properties, interpretation. Eur Respir J. 2010 Dec;36(6):1410-6. doi: 10.1183/09031936.00117509. Epub 2010 Jun 7. PMID 20530041
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Korn S, Both J, Jung M, Hubner M, Taube C, Buhl R. Prospective evaluation of current asthma control using ACQ and ACT compared with GINA criteria. Ann Allergy Asthma Immunol. 2011 Dec;107(6):474-9. doi: 10.1016/j.anai.2011.09.001. Epub 2011 Oct 5. PMID 22123375
- [Background] Schatz M, Sorkness CA, Li JT, Marcus P, Murray JJ, Nathan RA, Kosinski M, Pendergraft TB, Jhingran P. Asthma Control Test: reliability, validity, and responsiveness in patients not previously followed by asthma specialists. J Allergy Clin Immunol. 2006 Mar;117(3):549-56. doi: 10.1016/j.jaci.2006.01.011. PMID 16522452
- [Background] Thomas M, Kay S, Pike J, Williams A, Rosenzweig JR, Hillyer EV, Price D. The Asthma Control Test (ACT) as a predictor of GINA guideline-defined asthma control: analysis of a multinational cross-sectional survey. Prim Care Respir J. 2009 Mar;18(1):41-9. doi: 10.4104/pcrj.2009.00010. PMID 19240948
- [Background] Liu AH, Zeiger R, Sorkness C, Mahr T, Ostrom N, Burgess S, Rosenzweig JC, Manjunath R. Development and cross-sectional validation of the Childhood Asthma Control Test. J Allergy Clin Immunol. 2007 Apr;119(4):817-25. doi: 10.1016/j.jaci.2006.12.662. Epub 2007 Mar 13. PMID 17353040
- [Background] Liu AH, Zeiger RS, Sorkness CA, Ostrom NK, Chipps BE, Rosa K, Watson ME, Kaplan MS, Meurer JR, Mahr TA, Blaiss MS, Piault-Louis E, McDonald J. The Childhood Asthma Control Test: retrospective determination and clinical validation of a cut point to identify children with very poorly controlled asthma. J Allergy Clin Immunol. 2010 Aug;126(2):267-73, 273.e1. doi: 10.1016/j.jaci.2010.05.031. Epub 2010 Jul 10. PMID 20624640
- [Background] Juniper EF, Svensson K, Mork AC, Stahl E. Measurement properties and interpretation of three shortened versions of the asthma control questionnaire. Respir Med. 2005 May;99(5):553-8. doi: 10.1016/j.rmed.2004.10.008. Epub 2004 Nov 26. PMID 15823451
- [Background] Rhee H, Belyea MJ, Elward KS. Patterns of asthma control perception in adolescents: associations with psychosocial functioning. J Asthma. 2008 Sep;45(7):600-6. doi: 10.1080/02770900802126974. PMID 18773334
- [Background] Trochtenberg DS, BeLue R. Descriptors and perception of dyspnea in African-American asthmatics. J Asthma. 2007 Dec;44(10):811-5. doi: 10.1080/02770900701645769. PMID 18097855
- [Background] Trochtenberg DS, BeLue R, Piphus S, Washington N. Differing reports of asthma symptoms in African Americans and Caucasians. J Asthma. 2008 Mar;45(2):165-70. doi: 10.1080/02770900701847076. PMID 18350410
- [Background] Akinbami LJ, Moorman JE, Bailey C, Zahran HS, King M, Johnson CA, Liu X. Trends in asthma prevalence, health care use, and mortality in the United States, 2001-2010. NCHS Data Brief. 2012 May;(94):1-8. PMID 22617340
- [Background] Silvers SK, Lang DM. Asthma in African Americans: what can we do about the higher rates of disease? Cleve Clin J Med. 2012 Mar;79(3):193-201. doi: 10.3949/ccjm.79a.11016. PMID 22383554
- [Background] Haselkorn T, Lee JH, Mink DR, Weiss ST; TENOR Study Group. Racial disparities in asthma-related health outcomes in severe or difficult-to-treat asthma. Ann Allergy Asthma Immunol. 2008 Sep;101(3):256-63. doi: 10.1016/S1081-1206(10)60490-5. PMID 18814448
- [Background] Smith LA, Hatcher-Ross JL, Wertheimer R, Kahn RS. Rethinking race/ethnicity, income, and childhood asthma: racial/ethnic disparities concentrated among the very poor. Public Health Rep. 2005 Mar-Apr;120(2):109-16. doi: 10.1177/003335490512000203. PMID 15842111
- [Background] Leung TF, Tang NL, Wong GW, Fok TF. CD14 and toll-like receptors: potential contribution of genetic factors and mechanisms to inflammation and allergy. Curr Drug Targets Inflamm Allergy. 2005 Apr;4(2):169-75. doi: 10.2174/1568010053586336. PMID 15853738
- [Background] Okelo SO, Wu AW, Merriman B, Krishnan JA, Diette GB. Are physician estimates of asthma severity less accurate in black than in white patients? J Gen Intern Med. 2007 Jul;22(7):976-81. doi: 10.1007/s11606-007-0209-1. Epub 2007 Apr 24. PMID 17453263
- [Background] Velsor-Friedrich B, Militello LK, Richards MH, Harrison PR, Gross IM, Romero E, Bryant FB. Effects of coping-skills training in low-income urban African-American adolescents with asthma. J Asthma. 2012 May;49(4):372-9. doi: 10.3109/02770903.2012.660296. Epub 2012 Feb 21. PMID 22352813
- [Background] Leung TF, Ko FW, Sy HY, Wong E, Li CY, Yung E, Hui DS, Wong GW, Lai CK. Identifying uncontrolled asthma in young children: clinical scores or objective variables? J Asthma. 2009 Mar;46(2):130-5. doi: 10.1080/02770900802468533. PMID 19253117
- [Background] Koolen BB, Pijnenburg MW, Brackel HJ, Landstra AM, van den Berg NJ, Merkus PJ, Hop WC, Vaessen-Verberne AA. Comparing Global Initiative for Asthma (GINA) criteria with the Childhood Asthma Control Test (C-ACT) and Asthma Control Test (ACT). Eur Respir J. 2011 Sep;38(3):561-6. doi: 10.1183/09031936.00173710. Epub 2011 Mar 15. PMID 21406508
- [Background] Shi Y, Tatavoosian AV, Aledia AS, George SC, Galant SP. Cut points for Asthma Control Tests in Mexican children in Orange County, California. Ann Allergy Asthma Immunol. 2012 Aug;109(2):108-13. doi: 10.1016/j.anai.2012.06.002. Epub 2012 Jul 4. PMID 22840251
- [Background] Horak E, Grassl G, Skladal D, Ulmer H. Lung function and symptom perception in children with asthma and their parents. Pediatr Pulmonol. 2003 Jan;35(1):23-8. doi: 10.1002/ppul.10218. PMID 12461735
- [Background] Cabral AL, Conceicao GM, Saldiva PH, Martins MA. Effect of asthma severity on symptom perception in childhood asthma. Braz J Med Biol Res. 2002 Mar;35(3):319-27. doi: 10.1590/s0100-879x2002000300006. PMID 11887209
- [Background] Baker RR, Mishoe SC, Zaitoun FH, Arant CB, Lucas J, Rupp NT. Poor perception of airway obstruction in children with asthma. J Asthma. 2000;37(7):613-24. doi: 10.3109/02770900009090817. PMID 11059529
- [Background] Fritz GK, McQuaid EL, Kopel SJ, Seifer R, Klein RB, Mitchell DK, Esteban CA, Rodriguez-Santana J, Colon A, Alvarez M, Canino G. Ethnic differences in perception of lung function: a factor in pediatric asthma disparities? Am J Respir Crit Care Med. 2010 Jul 1;182(1):12-8. doi: 10.1164/rccm.200906-0836OC. Epub 2010 Mar 18. PMID 20299534
- [Background] Fritz GK, McQuaid EL, Spirito A, Klein RB. Symptom perception in pediatric asthma: relationship to functional morbidity and psychological factors. J Am Acad Child Adolesc Psychiatry. 1996 Aug;35(8):1033-41. doi: 10.1097/00004583-199608000-00014. PMID 8755800
- [Background] Mittal V, Khanna P, Panjabi C, Shah A. Subjective symptom perceptual accuracy in asthmatic children and their parents in India. Ann Allergy Asthma Immunol. 2006 Oct;97(4):484-9. doi: 10.1016/S1081-1206(10)60939-8. PMID 17069103
- [Background] Diette GB, Rand C. The contributing role of health-care communication to health disparities for minority patients with asthma. Chest. 2007 Nov;132(5 Suppl):802S-809S. doi: 10.1378/chest.07-1909. PMID 17998344
- [Background] Institute of Medicine (US) Committee on Health Literacy; Nielsen-Bohlman L, Panzer AM, Kindig DA, editors. Health Literacy: A Prescription to End Confusion. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK216032/ PMID 25009856
- [Background] Apter AJ, Cheng J, Small D, Bennett IM, Albert C, Fein DG, George M, Van Horne S. Asthma numeracy skill and health literacy. J Asthma. 2006 Nov;43(9):705-10. doi: 10.1080/02770900600925585. PMID 17092853
- [Background] Apter AJ, Paasche-Orlow MK, Remillard JT, Bennett IM, Ben-Joseph EP, Batista RM, Hyde J, Rudd RE. Numeracy and communication with patients: they are counting on us. J Gen Intern Med. 2008 Dec;23(12):2117-24. doi: 10.1007/s11606-008-0803-x. Epub 2008 Oct 2. PMID 18830764
- [Background] Jia CE, Zhang HP, Lv Y, Liang R, Jiang YQ, Powell H, Fu JJ, Wang L, Gibson PG, Wang G. The Asthma Control Test and Asthma Control Questionnaire for assessing asthma control: Systematic review and meta-analysis. J Allergy Clin Immunol. 2013 Mar;131(3):695-703. doi: 10.1016/j.jaci.2012.08.023. Epub 2012 Oct 8. PMID 23058645
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Derived] Burbank AJ, Todoric K, Steele P, Rosen J, Zhou H, Frye M, Loughlin CE, Ivins S, Mills K, Massey LD, Reeve BB, Hernandez ML. Age and African-American race impact the validity and reliability of the asthma control test in persistent asthmatics. Respir Res. 2018 Aug 15;19(1):152. doi: 10.1186/s12931-018-0858-0. PMID 30111326
- See also: Ethnic Disparitites in the Burden and Treatment of Asthma — http://www.aafa.org/media/Ethnic-Disparities-Burden-Treatment-Asthma-Report.pdf
- See also: American Lung Association; "State of Lung Disease in Diverse Communities 2010." www.lungusa.org; 2010; p1 — http://www.lungusa.org